CLINICAL TRIAL: NCT02590146
Title: Non-Pharmacologic Patient Centered Pain Control Adjuncts During First Trimester Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22893
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Pregnancy Termination; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Patients in this group will participate in pain management counseling and choose non-pharmacologic pain control supports to use during their procedure in addition to the standard of care pain management offered in the office
  Interventions: Behavioral: Non-pharmacologic pain control adjuncts
- Control group (No Intervention): Patients in this group will receive standard of care pain management offered in the office.

INTERVENTIONS:
Behavioral: Non-pharmacologic pain control adjuncts
  Arms: Intervention Group

SUMMARY:
This study will examine the use of non-pharmacologic pain control techniques and pain-management counseling as an additional tool for reducing pain during first trimester aspiration abortion.

ELIGIBILITY:
Inclusion Criteria:

* English speaking, able to read and understand consent form
* Age 18 + (minors eligible with parental consent)
* Seeking in-office aspiration termination of pregnancy
* Gestational age less than 14 weeks

Exclusion Criteria:

* Not able to read or understand English
* Unable to understand consent
* Minors without parental consent
* Requesting narcotic or sedative analgesics
* Currently incarcerated
* Gestational age greater than 14 weeks
* Seeking medication abortion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Difference in overall pain score during procedure between control and intervention group | Collected within 1 minute of procedure completion
  Patients will complete a visual analog scale to score their overall pain for the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hawaii, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No